CLINICAL TRIAL: NCT02866630
Title: Coronary Sinus Blood Sevoflurane and Desflurane Concentration and Lactate Changes in Patients Undergoing Heart Surgery
Acronym: SEVO-DES
Status: Withdrawn | Type: Observational
Why Stopped: No facility to measure volatile anaesthetic concentration in human blood sample
Sponsor: University of Malaya (Other)
Collaborators: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: UM-1
Record Dates: First submitted 2016-07-19; First posted 2016-08-15 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Myocardial Reperfusion Injury; Heart Diseases; Postoperative Complications
Keywords: Sevoflurane; Desflurane; Coronary Sinus; Oxygenator Exhaust; Lactate; Cardiopulmonary bypass
MeSH Terms: conditions — Myocardial Reperfusion Injury; Heart Diseases; Postoperative Complications | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cardiopulmonary bypass (Sevoflurane): All patients who scheduled for an elective heart surgery in University Malaya Medical Centre using a heart-lung machine and the administration of sevoflurane will be recruited in this study. The medical and surgical care plans for participants remain as usual in this study with an exception being six additional blood samples of about two-teaspoonful in volume will be collected from an in-placed catheters in vein and aorta.
  Interventions: Biological: Blood samples
- Cardiopulmonary bypass (Desflurane): All patients who scheduled for an elective heart surgery in University Malaya Medical Centre using a heart-lung machine and the administration of desflurane will be recruited in this study. The medical and surgical care plans for participants remain as usual in this study with an exception being six additional blood samples of about two-teaspoonful in volume will be collected from an in-placed catheters in vein and aorta.
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — Six additional blood samples will be taken from in-situ catheters during heart surgery

SUMMARY:
In the last few years, anaesthetics gas such as isoflurane, desflurane and sevoflurane used in heart surgery have shown some benefits to reduce the risk of heart muscle damage than total intravenous anesthetics. A study by the investigators suggested that isoflurane needs a longer duration to achieve equilibrium between coronary sinus and radial artery, indicating that isoflurane in coronary sinus does not accurately reflect its level in the heart muscle. Different agents have unique characteristics with different equilibration rate. However, the levels of sevoflurane and desflurane in coronary sinus and radial artery have not been measured. In addition, lactate is believed to be a very useful indicator to predict the outcome of recovery phase after any surgery. This study aims to measure the level of sevoflurane or desflurane in blood circulation. It will also assess whether sevoflurane or desflurane concentration in the blood is correlated to the its oxygenator exhaust level and affected by temperature, haematocrit level and gas flow rate during heart-lung machine. It also aims to examine the association of lactate and the outcomes of cardiac patient in intensive care unit after cardiac surgery.

DETAILED DESCRIPTION:
In recent years, many clinical trials have demonstrated the myocardial protective properties of volatile anaesthetic agent through a similar mechanism as ischaemic pre-conditioning. It is hypothesised that volatile anaesthetic agent promotes the generation of nitric oxide and reactive oxygen species, which then activates the adenosine receptor, and subsequently initiates the opening of mitochondrial potassium ion channel to minimise perioperative myocardial injury. Many researchers have studied the protective benefit of volatile anaesthesia in heart surgery that involves CPB machine over the last 10 years. In 2006, a meta-analysis of 27 clinical trials have demonstrated that patients receiving volatile anaesthesia either isoflurane, sevoflurane, desflurane or enflurane, experienced lesser myocardial injury, required shorter duration of mechanical ventilation and shorter hospital stay as compared to those tranquilised with a total intravenous anaesthesia technique.

In the administration of volatile anaesthetic agent, the literature review of optimal dosing and timing are not clinically well-established. Unpublished data from the investigators shows that isoflurane requires slightly longer duration to achieve equilibrium between coronary sinus and radial artery, indicating that coronary sinus isoflurane concentration does not accurately reflect its level in myocardium. Also, the temperature of CPB, haematocrit level and gas flow rate appeared to affect the plasma isoflurane concentration to a certain extent. In addition, the investigators only managed to look at isoflurane itself, where other types of volatile anaesthetics namely sevoflurane and desflurane have different nature characteristics and possibly yield to different findings. Furthermore, lactate is believed to be a useful indicator for the outcome of recovery post-operatively. However, it remains unknown that whether would the lactate levels change significantly before, during and after cardiac surgery.

Theoretically, the measurement of volatile anaesthetics concentration in the heart would require a biopsy of heart muscle. Able to identify the level of myocardial anaesthetic level from coronary sinus could be a non-invasive measurement for future studies to look at the optimal concentrations of volatile anaesthetics required to achieve its pharmacological ischaemic pre-conditioning to minimise myocardial damage perioperatively.

The main aim of this study is to determine the level of myocardial sevoflurane or desflurane concentration from coronary sinus blood sample that taken from a coronary sinus catheter, which is routinely inserted to administer retrograde cardioplegia solution instead of invasive biopsy method. This study will also examine the association between the coronary sinus sevoflurane or desflurane concentration and its oxygenator exhaust level during CPB and investigate the influence of temperature, gas flow rate and haematocrit level on plasma sevoflurane or desflurane concentrations. A secondary analysis aims to determine the changes of lactate levels before, during and after cardiac surgery, and the recovery outcomes of cardiac patients in intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Scheduled for elective cardiac surgery.
* Anaesthetised using sevoflurane or desflurane throughout the whole operation
* Patient has consented to participate

Exclusion Criteria:

* Emergency surgery or patient with malignancy
* Heart surgery undertaken without CPB
* Age younger than 18 years
* Unable or unwilling to provide informed consent
* Anaesthetised using total intravenous-based technique

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who scheduled for an elective heart surgery in University Malaya Medical Centre involving the administration of sevoflurane or desflurane throughout the operation will be recruited in this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-07-20 (Estimated); Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The Concentration of Anaesthetics in Coronary Sinus and Radial Arterial | 1 weeks after blood samples taken
  All blood samples will be analysed twice for sevoflurane or desflurane with a high performance gas chromatography and mass spectrometry detector (Thermo Scientific TSQ Ultra Triple Quadrupole GC-MS) with a Headspace Autosampler (TriPlus 300). Blood samples were quantified using an external calibration curve prepared in a controlled whole blood over a range of sevoflurane or desflurane concentrations. The reporting measurement unit for sevoflurane or desflurane concentration will be μgmL-1.

SECONDARY OUTCOMES:
Oxygenator exhaust sevoflurane or desflurane levels on heart-lung machine | 1 week after measurement of oxygenator exhaust isoflurane gas
  The measurement unit for oxygenator exhaust anaesthesia level will be in %, which is analysed by an infrared anaesthetic gas analyser.
Lactate levels before and after surgery | Lactate measurement at 30 mins before and 1 hour after cardiac surgery
  The measurement for lactate level will be in mmolL-1, which is analysed by lactate testing equipment in theatre.

CONTACTS AND LOCATIONS:
Overall Officials: Chew Yin Wang, FRCA (Eng), Principal Investigator — University of Malaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belhomme D, Peynet J, Louzy M, Launay JM, Kitakaze M, Menasche P. Evidence for preconditioning by isoflurane in coronary artery bypass graft surgery. Circulation. 1999 Nov 9;100(19 Suppl):II340-4. doi: 10.1161/01.cir.100.suppl_2.ii-340. PMID 10567326
- [Background] Landoni G, Greco T, Biondi-Zoccai G, Nigro Neto C, Febres D, Pintaudi M, Pasin L, Cabrini L, Finco G, Zangrillo A. Anaesthetic drugs and survival: a Bayesian network meta-analysis of randomized trials in cardiac surgery. Br J Anaesth. 2013 Dec;111(6):886-96. doi: 10.1093/bja/aet231. Epub 2013 Jul 12. PMID 23852263
- [Background] Marco R. Cardiopulmonary bypass. In: Alston, RP, Myles, PS, Ranucci M, editor. Oxford Textbook of Cardiothoracic Anaesthesia. 1st ed. Oxford: Oxford University Press; 2015. p. 117-30.
- [Background] Pramood, CK, Reena, S, Gajraj S. Ischemic and anesthetic preconditioning of the heart: an insight into the concepts and mechanisms. J Indian Acad Clin Med. 2005;6(1):45-7.
- [Background] Yoshimi I. Cardiac preconditioning by anesthetic agents: roles of volatile anesthetics and opioids in cardioprotection. Yonago Acta Med. 2007;50:45-55.
- [Background] Irwin, Michael G, Wong GT. Myocardial Protection During Cardiac Surgery. In: Alston, R Peter, Myles, Paul S, Ranucci M, editor. Oxford Textbook of Cardiothoracic Anaesthesia. 1st ed. Oxford: Oxford University Press; 2015. p. 157-63.
- [Background] Symons JA, Myles PS. Myocardial protection with volatile anaesthetic agents during coronary artery bypass surgery: a meta-analysis. Br J Anaesth. 2006 Aug;97(2):127-36. doi: 10.1093/bja/ael149. Epub 2006 Jun 21. PMID 16793778
- [Background] Ng, KT, Alston, P. The Levels of Anaesthetics in Heart Muscle During Heart Surgery (TLAHMHS) [Internet]. ClinicalTrial.gov.my. 2015. Available from: https://clinicaltrials.gov/ct2/show/NCT02471001